CLINICAL TRIAL: NCT02345343
Title: Early Post-Marketing Study of Eliquis (Apixaban), in Treatment of Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE), and Prevention of Recurrent DVT and PE in Adults
Brief Title: Early Post-Marketing Study of ELIQUIS (Apixaban) in Mexico
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-399
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug: Apixaban: Patients with VTE who are being given apixaban for the treatment and/or prevention of recurrence of DVT and PE at the sentinel site
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis

SUMMARY:
The primary objective of the study is to report adverse events of on-treatment AEs by the treating physicians during a specified 24-month study period in patients with venous thromboembolism at the sentinel site(s) for the National Center of Pharmacovigilance (CNFV) in Mexico.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients 18 years old with DVT and PE at the sentinel site who received at least 1 dose of apixaban for the treatment and/or prevention of recurrence of DVT and PE during the specified 24-month study period

Exclusion Criteria:

* Subjects who received apixaban as part of a clinical trial
* Subjects who received apixaban for any indication other than local approved
* Contraindications included in the approved Mexican prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sentinel site for the CNFV in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05-04 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
The number of adverse events (AEs) notified to health authorities (HAs) of on-treatment AEs by the treating physicians | Up to 24-month study period

SECONDARY OUTCOMES:
The AEs reported to HA in a table format identifying the report number, patient ID number, and type of AE | Up to 24-month study period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Querétaro, Mexico

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx